CLINICAL TRIAL: NCT02104284
Title: A Comparative Bronchial Provocation Study With Mannitol and Methacolinie in a Korean Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BL&H Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: mannitol-01
Record Dates: First submitted 2014-03-21; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-04

CONDITIONS: Asthma
Keywords: Bronchial provocation test; Mannitol; Methacholine; Bronchial hyperreactivity; Sensitivity and specificity
MeSH Terms: conditions — Asthma; Bronchial Hyperreactivity; Hypersensitivity | interventions — Methacholine Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Normal controls, methacholine positive (Other): methacholine and mannitol bronchial challenge tests: Positive methacholine challenge tests in normal controls
  Interventions: Procedure: methacholine and mannitol bronchial challenge tests
- Normal controls, mannitol (Other): methacholine and mannitol bronchial challenge tests: Positive mannitol challenge tests in normal controls.
  Interventions: Procedure: methacholine and mannitol bronchial challenge tests
- Asthma, Methacholine (Active Comparator): methacholine and mannitol bronchial challenge tests: Positive methacholine challenge tests in asthmatics
  Interventions: Procedure: methacholine and mannitol bronchial challenge tests
- Asthma, Mannitol (Active Comparator): methacholine and mannitol bronchial challenge tests: Positive mannitol challenge tests in asthmatics
  Interventions: Procedure: methacholine and mannitol bronchial challenge tests

INTERVENTIONS:
Procedure: methacholine and mannitol bronchial challenge tests — Airway hyperresponsiveness is a common feature of asthma. Methacholine and mannitol are two representative agonists for bronchial challenge. They have theoretically different mechanisms of action, and may have different diagnostic properties. However, their difference has not been directly evaluated among Korean adults. In this study, we compare the diagnostic properties of methacholine and mannitol bronchial provocation tests.
  Asthmatic patients and non-asthmatic controls were recruited prospectively from four referral hospitals in Korea. Participants were challenged with each of methacholine and mannitol inhalation on different days. Their diagnostic utility was evaluated by calculating their sensitivity, specificity, positive/negative predictive values for asthma diagnosis.

SUMMARY:
Asthmatic patients and non-asthmatic controls were recruited prospectively from four referral hospitals in Korea. Participants were challenged with each of methacholine and mannitol inhalation on different days. Their diagnostic utility was evaluated by calculating their sensitivity and specificity for asthma diagnosis. Response-dose-ratio was also compared.

DETAILED DESCRIPTION:
This study was a prospective, multicenter study performed at four referral hospitals in Korea: Seoul National University Hospital, Samsung Medical Center, Ajou University Hospital, and Hanyang University Medical Center. Hospital-based recruitment was performed for asthmatic patients and non-asthmatic controls. Asthmatic patients were defined as those who had been diagnosed with asthma by specialist physicians; they had recurrent symptoms of asthma (wheezing and dyspnea) and used anti-asthmatic medication for 6 months before the enrollment. Non-asthmatic controls were voluntarily recruited from hospital visitors; they were included if they had never wheeze or physician diagnosed asthma.

Common inclusion criteria were Korean adults between the age of 18 and 70 years who could understand and perform lung function tests and bronchial challenges. Exclusion criteria were any one of following: history of recent respiratory infection (within the last 4 weeks), history of a recent surgery, history of heart disease that could impose risks during bronchial challenges, history of uncontrolled hypertension, current smokers or ex-smokers with more than 10 pack-years, history of known pulmonary diseases with the exception of asthma, pregnancy or lactation, severe obesity (body mass index [BMI] of >35 kg/m2), history of any health condition considered inappropriate for participation in this study, or a pre-bronchodilator predictive value of forced expiratory volume in 1 second (FEV1) of <70%.

All participants underwent methacholine bronchial challenge test and mannitol challenge test on different days, separated by least 24 h, as in previous reports.7, 10 All asthmatic patients stopped their anti-asthma medications before the tests according to the predetermined protocols. The protocol was approved by the Institutional Review Board of Seoul National University Hospital. All subjects gave written informed consent.

Methacholine challenge test> The methacholine challenge test was performed as previously described.11, 12 Pulmonary function testing was carried out using a spirometry system (SensorMedics 2130; SensorMedics, CA, USA). The methacholine challenge test was performed using the Chai method13 with minor modifications. Briefly, methacholine was prepared at the following concentrations, diluted with saline: 0.25, 0.625, 1, 4, 16, and 25 mg/mL. Methacholine was delivered as an aerosol by a Rosenthal-French dosimeter (Laboratory for Applied Immunology, Inc., Baltimore, MD) and a nebulizer. Subjects were instructed to inhale five inspiratory capacity breaths while increasing the methacholine concentration from 0.25 to 25 mg/mL. The methacholine concentration that caused a 20% decrease in the FEV1 from baseline was defined as PC20. AHR was defined as positive at PC20 < 16 mg/mL.

Mannitol challenge test> A commercial mannitol (Aridol™; BL&H Co., Ltd., South Korea) kit was used, and the challenge test was performed according to the manufacturer's protocols.14 The mannitol capsule dose started at 0 mg and increased to a total cumulative dose of 635 mg. Each capsule was placed in the inhalation device, and a hole was made by pressing the device button before inhalation. After a deep breath of mannitol, the FEV1 was measured after 60 seconds. The test was considered positive if the FEV1 value decreased by more than 15% compared with the baseline FEV1. The cumulative mannitol dose that caused a 15% decrease in the FEV1 from baseline was defined as PD15. If the FEV1 did not decline by more than 15%, the dose was increased until a cumulative dose of 635 mg was reached. If the FEV1 did not fall by more than 15% until the last dose, the test was considered negative.

ELIGIBILITY:
Inclusion Criteria:

* Common inclusion criteria were Korean adults between the age of 18 and 70 years who could understand and perform lung function tests and bronchial challenges.

Exclusion Criteria:

* History of recent respiratory infection (within the last 4 weeks)
* History of a recent surgery
* History of heart disease that could impose risks during bronchial challenges
* History of uncontrolled hypertension
* Current smokers or ex-smokers with more than 10 pack-years
* History of known pulmonary diseases with the exception of asthma
* Pregnancy or lactation
* Severe obesity (body mass index [BMI] of >35 kg/m2)
* History of any health condition considered inappropriate for participation in this study
* Pre-bronchodilator predictive value of forced expiratory volume in 1 second (FEV1) of <70%

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
sensitivity comparison of the mannitol challenge test and methacholine challenge test | 60 minutes
  The diagnostic properties of the mannitol challenge test and methacholine challenge test (sensitivity, specificity, positive predictive value, and negative predictive value) were calculated against the physician's diagnosis of asthma.
  methacholine challenge test: positive at PC20 < 16 mg/mL mannitoln test: positive if FEV1 fell by more than 15% until the last dose (until a cumulative dose of 635 mg) gold standard: physician's diagnosis of asthma
  sensitivity: true positive / true positive+false negative

SECONDARY OUTCOMES:
specificity comparison of the mannitol challenge test and methacholine challenge test | 60 minutes
  The diagnostic properties of the mannitol challenge test and methacholine challenge test (sensitivity, specificity, positive predictive value, and negative predictive value) were calculated against the physician's diagnosis of asthma.
  methacholine challenge test: positive at PC20 < 16 mg/mL mannitoln test: positive if FEV1 fell by more than 15% until the last dose (until a cumulative dose of 635 mg) gold standard: physician's diagnosis of asthma
  specificity: true negative / false positive+true negative
positive predictive value comparison of the mannitol challenge test and methacholine challenge test | 60 minutes
  The diagnostic properties of the mannitol challenge test and methacholine challenge test (sensitivity, specificity, positive predictive value, and negative predictive value) were calculated against the physician's diagnosis of asthma.
  methacholine challenge test: positive at PC20 < 16 mg/mL mannitoln test: positive if FEV1 fell by more than 15% until the last dose (until a cumulative dose of 635 mg) gold standard: physician's diagnosis of asthma
  positive predictive value: true positive / true positive+false positive
negative predictive value comparison of the mannitol challenge test and methacholine challenge test | 60 minutes
  The diagnostic properties of the mannitol challenge test and methacholine challenge test (sensitivity, specificity, positive predictive value, and negative predictive value) were calculated against the physician's diagnosis of asthma.
  methacholine challenge test: positive at PC20 < 16 mg/mL mannitoln test: positive if FEV1 fell by more than 15% until the last dose (until a cumulative dose of 635 mg) gold standard: physician's diagnosis of asthma
  negative predictive value: true negative / true negative+false negative

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Heon Cho, M.D.,Ph.D., Principal Investigator — Seoul National University College of Medicine

REFERENCES:
- [Derived] Kim MH, Song WJ, Kim TW, Jin HJ, Sin YS, Ye YM, Kim SH, Park HW, Lee BJ, Park HS, Yoon HJ, Choi DC, Min KU, Cho SH. Diagnostic properties of the methacholine and mannitol bronchial challenge tests: a comparison study. Respirology. 2014 Aug;19(6):852-6. doi: 10.1111/resp.12334. Epub 2014 Jun 26. PMID 24975800